CLINICAL TRIAL: NCT00206921
Title: Pulsed Dye Laser and Intense Pulsed Light for the Treatment of Telangiectasia and Skin Redness
Brief Title: Pulsed Dye Laser and Intense Pulsed Light (IPL) for the Treatment of Telangiectasia and Skin Redness
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bispebjerg Hospital (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: KF-01-236/04
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2007-07-25 (Estimated); Status verified 2004-12

CONDITIONS: Telangiectasis; Erythema
Keywords: Telangiectasia; Skin redness
MeSH Terms: conditions — Telangiectasis; Erythema | interventions — Lasers, Dye; Intense Pulsed Light Therapy

INTERVENTIONS:
Device: Pulsed dye laser
Device: Intense pulsed light

SUMMARY:
The purpose of the study is to compare efficacy and adverse effects of pulsed dye laser and intense pulsed light in patients with skin telangiectasia and redness.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Skin types I, II, III
* No previous laser or IPL treatment for the condition

Exclusion Criteria:

* Younger than 18 years old
* Skin types IV, V, or VI
* Pregnant or lactating women
* Previous laser or IPL treatment for the condition
* Recent exposure to sun or sun-beds
* Treatment with oral retinoid within 6 months
* Tendency to produce hypertrophic scars or keloids

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2005-02; Study Completion 2005-08

CONTACTS AND LOCATIONS:
Overall Officials: Merete Hædersdal, MD, PhD, DrMedSci, Principal Investigator — Bispebjerg Hospital
Locations (1):
- Bispebjerg Hospital, Copenhagen, Copenhagen NV, Denmark